CLINICAL TRIAL: NCT02434926
Title: Anesthetic Management in Fetoscopic Surgery and Incidence of Complications - A Retrospective Review
Brief Title: Anesthetic Management in Fetoscopic Surgery and Incidence of Complications
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 150/2558(EC2)
Record Dates: First submitted 2015-04-26; First posted 2015-05-06 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Fetoscopy; Anesthetic Complications; Pregnancy
Keywords: fetoscopy; fetal surgery; anesthetic complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Fetoscopic surgery has been acknowledged to be a reliable procedure to correct several congenital anomalies e.g. shunt insertion in fetal bladder outlet obstruction, laser ablation of vessels in twin-twin transfusion syndrome (TTTS), balloon occlusion in congenital diaphragmatic hernia etc. The technique involves an introduction of small-caliber instruments into the amniotic cavity under ultrasound guidance. This procedure can be successfully done under either general anesthesia, regional anesthesia or local anesthesia with sedation. Each technique has both advantages and drawbacks.

Several complications related to anesthetic after fetoscopic surgery can occur. For instance, pulmonary edema which is caused by intravenous fluid loading, irrigation fluid absorption or fluid flow through myometrium venous channel. Besides, maternal hypotension intraoperatively can arise from spinal anesthesia.

The aim of the study is to report choice of anesthesia using in fetoscopic surgery in the tertiary care institute (Siriraj hospital) and incidence of complications which may relate to different anesthetic techniques.

DETAILED DESCRIPTION:
The quantity and types of medications using in different anesthetic technique will be gathered including opioid, benzodiazepine, propofol, detail of drugs making fetal paralysis, amount of local anesthetic drug in spinal anesthesia etc. Tocolytic drug will also be recorded eg. terbutaline, nifedipine or magnesium sulfate. These drugs have been generally known that may cause hypotension or pulmonary edema.

In intraoperative period, the investigators emphasize in the incidence of hypotension and other possible complications such as pulmonary aspiration, failed intubation, maternal desaturation or maternal bradycardia. Volume of intravenous fluid administered and amount of irrigation fluid will also be recorded.

Maternal and fetal outcome in recovery room and in postoperative period will be collected.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women who received intrauterine minimally invasive surgery from the past until 30 Nov 2015

Exclusion Criteria:

* pregnant women who received intrauterine minimally invasive surgery which was not anesthetized by anesthesiologist.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women who received fetocsopic surgery for any reasons eg. laser ablation of vessels in twin-twin transfusion syndrome, balloon occlusion in fetal congenital diaphragmatic hernia, fetal bladder outlet obstruction, intrauterine blood transfusion etc.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Type of anesthetic techniques used in fetoscopic surgery | in operating theatre
  Type of anesthetic techniques eg. general anesthesia, regional anesthesia, local anesthesia with sedation.

SECONDARY OUTCOMES:
Types and quantity of anesthetic medications used | in operating theatre
  Types and quantity of anesthetic medications used for anesthetize patients in different anesthetic techniques.
Incidence of complications | in operating theatre
  Intraoperative complications eg. failed intubation, aspiration, hypotension from spinal anesthesia, high spinal block, desaturation etc.
Incidence of complications | after surgery till patients discharge from the hospital
  Complications occurring postoperatively include pulmonary edema, fatal death etc.

CONTACTS AND LOCATIONS:
Overall Officials: Patchareya Nivatpumin, M.D., Principal Investigator — Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand
Locations (2):
- Thailand (2):
  - Anesthesiology department, Siriraj hospital, Mahidol University, Bangkok
  - Siriraj Hospital, Mahidol University, Bangkok

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nivatpumin P, Pangthipampai P, Jirativanont T, Dej-Arkom S, Triyasunant N, Tempeetikul T. Anesthetic Techniques and Incidence of Complications in Fetoscopic Surgery. J Med Assoc Thai. 2016 May;99(5):602-10. PMID 27501618